CLINICAL TRIAL: NCT05636722
Title: Evaluation of an Unguided Web-based Intervention for Students With Suicidal Ideation
Brief Title: Online Self-help for Students With Suicidal Ideation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. Technical reasons with the online platform for students.
  2. Limited number of students using the modules of self-help for suicide: recruitment was not started and the study was withdrawn.
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/BC-11287
Record Dates: First submitted 2022-11-08; First posted 2022-12-05 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants in this group (all participants) were asked to complete a questionnaire before and after (6 weeks after baseline) using the online self-help intervention (unguided web-based intervention).
  Interventions: Behavioral: Unguided web-based intervention

INTERVENTIONS:
Behavioral: Unguided web-based intervention — An online unguided intervention based on Cognitive Behavioural Therapy and elements of Dialectical Behaviour Therapy, Problem Solving Therapy, and Mindfulness Based Cognitive Therapy. The intervention consists of 6 modules with each a theoretical part, a weekly assignment and (optional and mandatory) exercises. Participants are advised to complete one module weekly. The original intervention was adapted to students (language, addition of podcasts, examples that were more suited to their lives).

SUMMARY:
The main goal of this study is to evaluate the effectiveness of an unguided web-based intervention for (college/university) students with suicidal ideation. This study will test the effectiveness by studying the effect on suicidal ideation and related outcomes (hopelessness and worrying) through a pre-post study design.

ELIGIBILITY:
Inclusion Criteria:

* Be student at a university or college
* Have suicidal thoughts
* ≥ 18 years old
* Have access to internet and a computer/laptop/smartphone
* Speak Dutch

Exclusion Criteria:

* /

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation: Beck Scale for Suicide Ideation | Baseline (right before the intervention)
  A 21-item self-report questionnaire to measure (the severity of) suicidal ideation in adolescents and adults. Each item is rated on a scale from 0 to 2, resulting in a total score ranging from 0 to 38, with higher scores indicating more (severe) suicidal ideation.
Suicidal ideation: Beck Scale for Suicide Ideation | posttest (6 weeks after baseline)
  A 21-item self-report questionnaire to measure (the severity of) suicidal ideation in adolescents and adults. Each item is rated on a scale from 0 to 2, resulting in a total score ranging from 0 to 38, with higher scores indicating more (severe) suicidal ideation.

SECONDARY OUTCOMES:
Hopelessness: The Beck Hopelessness Scale, 4-item version | Baseline (right before the intervention)
  A 4-item self-report questionnaire to measure hopelessness in adolescents and adults. Each item is rated as 'true' (score = 1) or 'false' (score = 0) for them over the past week, resulting in a total score ranging from 0 to 4, with higher scores indicating higher levels of hopelessness.
Hopelessness: The Beck Hopelessness Scale, 4-item version | posttest (6 weeks after baseline)
  A 4-item self-report questionnaire to measure hopelessness in adolescents and adults. Each item is rated as 'true' (score = 1) or 'false' (score = 0) for them over the past week, resulting in a total score ranging from 0 to 4, with higher scores indicating higher levels of hopelessness.
Worrying: Penn State Worry Questionnaire Past Week | Baseline (right before the intervention)
  A 15-item self-report questionnaire to measure worrying in the past week. Each item is rated on a 7-point Likert scale ranging from 0 ("never") to 6 ("almost always").
Worrying: Penn State Worry Questionnaire Past Week | posttest (6 weeks after baseline)
  A 15-item self-report questionnaire to measure worrying in the past week. Each item is rated on a 7-point Likert scale ranging from 0 ("never") to 6 ("almost always").

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Phd, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No